CLINICAL TRIAL: NCT03962348
Title: Reducing Duration of Untreated Psychosis Through Early Detection in a Large Jail System - Clinical Interviews With Detainees With Early Psychosis
Brief Title: Clinical Interviews With Detainees With Early Psychosis
Acronym: Interview
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Vera Institute of Justice (Other); University of Illinois at Chicago (Other); University of South Florida (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Michael Compton, Professor of Psychiatry, Columbia University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: NYSPI 7771 - 251051; R34MH117766 (NIH)
Record Dates: First submitted 2019-05-19; First posted 2019-05-24 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: First-Episode Psychosis
Keywords: Detainees; Early Psychosis
MeSH Terms: conditions — Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: Feasibility and Acceptability Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Specialized Early Engagement Support Service (Experimental): The investigators will implement a Specialized Early Engagement Support Service (SEESS) in the same three jails. The SEESS will increase the likelihood that referred individuals found to have first-episode psychosis enroll in Coordinated Specialty Care upon release.
  Interventions: Behavioral: Specialized Early Engagement Support Service

INTERVENTIONS:
Behavioral: Specialized Early Engagement Support Service — The Specialized Early Engagement Support Service (SEESS - a Social Worker and Peer Specialist) will link detainees with first-episode psychosis (FEP), using tenets of person-centered treatment and shared decision-making, and the Critical Time Intervention model, to community-based Coordinated Specialty Care (CSC).

SUMMARY:
The investigators are studying a jail-based intervention to reduce the duration of untreated psychosis (DUP) among young adults with previously undetected first-episode psychosis who are detained in jail. Longer DUP (or treatment delay) is linked to poorer outcomes in first-episode psychosis and there is evidence that justice-involved young adults with first-episode psychosis have an alarmingly long DUP. Thus, despite the expansion of Coordinated Specialty Care (CSC) programs that improve outcomes through early, multi-component care, there is a need to establish early detection services in the criminal justice system and create pathways from justice involvement to CSC. This intervention offers a novel and potentially high impact approach for reducing DUP in jail settings: a jail-based Specialized Early Engagement Support Service that receives referrals, engages detainees, and serves as a bridge to community-based CSC. The study team will design and implement the intervention, thoroughly study its feasibility and acceptability, and prepare an intervention manual for broader use in diverse jails and future formal research.

DETAILED DESCRIPTION:
Persons with serious mental illnesses are overrepresented in jails. Criminal justice (CJ) involvement, including jail detention, is common among those with first-episode psychosis (FEP) and frequently precedes psychiatric treatment engagement. Yet, no documented interventions currently exist specifically to identify/engage such individuals while in jail and connect them to Coordinated Specialty Care (CSC) in the community upon release. Expansion of CSC programs across the U.S. provides an opportunity for partnership with the CJ system-one that has the potential to reduce the duration of untreated psychosis (DUP) and thus improve outcomes.

To detect FEP and reduce DUP among detainees in a large, urban jail, the investigators propose to implement: a Specialized Early Engagement Support Service (SEESS) in 3 jails on Rikers Island in New York City (NYC): Anna M. Kross Center (AMKC), Rose M. Singer Center (RMSC) and Robert N. Davoren Complex (RNDC).

The investigators expect the multimedia TEC to generate referrals to the Correctional Health Services (CHS), and to reduce DUP-1 (psychosis onset to antipsychotic initiation). Then, the jail-based SEESS (a Social Worker and Peer Specialist) will link those identified to community-based CSC (primarily OnTrackNY sites in NYC), thus reducing DUP-2 (psychosis onset to CSC enrollment).

The investigators will examine a set of hypothesized targets/mediators (the "how's"). These are key ingredients that underpin the intervention's ability to reduce DUP.

The multi-media TEC will generate referrals to the CHS, by improving the behavioral capabilities, expectations, and self-efficacy (constructs from Social Cognitive Theory) of the Correction Officers trained. The SEESS will then link detainees with FEP, using tenets of person-centered treatment and shared decision-making, and the Critical Time Intervention model, to community-based CSC. This will occur through engagement of detainees while in jail, and telephonically (when possible) after release. The investigators will assess feasibility and acceptability to lay the groundwork for a multi-site, definitive effectiveness trial.

ELIGIBILITY:
Inclusion Criteria:

* Detainees that have been referred by Correctional Health Services as experiencing early-course or first-episode psychosis
* between the ages of 18 and 30 years
* have a Mini-Mental State Examination (MMSE) score of >23
* have the capacity to provide informed consent for the study
* able to understand and speak English

Exclusion Criteria:

* children under the age of 18 years

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-01-08 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2023-03-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Compton, MD, MPH, Principal Investigator — Columbia University
Locations (1):
- Rikers Island Jails (Anna M. Kross Center, Rose M. Singer Center, and Robert N. Davoren Complex), East Elmhurst, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected from this clinical trials research will be deposited into the National Institute of Mental Health Data Archive (NDA). In order to deposit the data, the investigators will use a consent form that allows broad data sharing within the research community. A global unique identifier (GUID) will be created for each research participant using the software that NIMH will provide. Dr. Compton and the research coordinator will work with NIMH to create data dictionaries that are relevant to their research. The investigators will share our results, positive and negative, specific to the cohorts and outcome measures studied
Time Frame: To be determined
Access Criteria: To be determined

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Specialized Early Engagement Support Service
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Specialized Early Engagement Support Service
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 22.75 [18 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Black or African American | 6
  Race: White or Caucasian | 0
  Race: Asian | 0
  Race: American Indian or Alaska Native | 0
  Race: Native Hawaiian or other Pacific Islander | 0
  Race: Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Referrals to Correctional Health Services (CHS)
Description: This primary measure reports the numbers of referrals of detainees with early psychosis from the Rikers project.
Time Frame: 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Specialized Early Engagement Support Service
Number analyzed (Participants) | 8
Participants | 8

2. Primary Outcome: Number of Referrals to Coordinated Specialty Care (CSC)
Description: Number individuals found to have first-episode psychosis enrolled in CSC upon release from jail.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Specialized Early Engagement Support Service
Number analyzed (Participants) | 8
Participants | 1

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Specialized Early Engagement Support Service
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
This was a very small study, and statistical analyses were therefore not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT03962348/Prot_001.pdf
  • Informed Consent Form (2019-05-13): https://cdn.clinicaltrials.gov/large-docs/48/NCT03962348/ICF_000.pdf